CLINICAL TRIAL: NCT05961800
Title: OMEGA Study: Offset Mechanisms in Evaluation of Lumbar Medial Branch Block
Brief Title: Offset Mechanisms in Evaluation of Lumbar Medial Branch Blocks
Acronym: OMEGA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Benedict Alter, Assistant Professor, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY23040122
Record Dates: First submitted 2023-07-05; First posted 2023-07-27 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Pain, Chronic; Facet Joint Pain; Pain, Procedural; Analgesia
Keywords: lumbar; medial branch block; offset analgesia; onset hyperalgesia; QST; quantitative sensory testing
MeSH Terms: conditions — Chronic Pain; Pain, Procedural; Agnosia

STUDY DESIGN:
Intervention Model Description: Quantitative Sensory Testing
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Quantitative Sensory Testing (Experimental): Participants with chronic low back pain and a scheduled lumbar medial branch block undergo quantitative sensory testing.
  Interventions: Behavioral: Cutaneous Probe; Behavioral: Quantitative Sensory Testing; Behavioral: Computer Tasks

INTERVENTIONS:
Behavioral: Cutaneous Probe — A computer-controlled probe delivers temperatures to the skin to measure pain, offset analgesia and onset hyperalgesia.
Behavioral: Quantitative Sensory Testing — Standard methods involving pinprick, pressure, heat, and cold applied to the skin are used to measure sensation and pain
Behavioral: Computer Tasks — Quantitative Sensory Testing (QST) and computer tasks are used to measure changes in pain intensity.

SUMMARY:
This study examines the relationship between central nervous system (CNS) mechanisms of pain inhibition and the pain relief that occurs following a lumbar medial branch block (MBB).

DETAILED DESCRIPTION:
This study examines the relationship between central nervous system (CNS) mechanisms of pain inhibition and the pain relief that occurs following a commonly-performed nerve block used to diagnose and treat chronic low back pain. Patients scheduled for lumbar medial branch blocks as part of routine clinical care will arrive to clinic prior to the block for quantitative sensory testing procedures that measure CNS pain modulation. Patients will then undergo treatment as usual with their block, subsequently reporting low back pain intensity in a pain diary.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for lumbar MBB in UPMC Pain Management clinics
* Age > 18 years old
* Predominantly axial chronic low back pain at least 3 months on a daily basis
* Must meet the minimum criteria for cognitive function using the PROMIS 2-item cognitive screener (>3)
* Low back pain intensity of > 3/10
* Willing and able to receive study-related phone calls

Exclusion Criteria:

* History of spine surgery at the level of the lumbar MBB
* Active worker's compensation or litigation claims
* New pain and/or psychiatric treatments within 2 weeks of enrollment
* Not fluent in English and/or not able to complete the questionnaires
* Any clinically unstable systemic illness that is judged to interfere with the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-07-05 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Offset analgesia and onset hyperalgesia | during this portion of the study visit (30 minutes)
  Pain intensity difference during heat stimuli measured on a 0-100 sliding scale (0 is no pain, 100 is the most intense pain imaginable) at baseline
Low back pain intensity change | Immediately after lumbar medial branch block and up to 16 hours after lumbar medial branch block
  Patients respond to the question "How would you rate your back pain right now?" from 0 (no pain) to 10 (worst imaginable pain) to see how intense their back pain is each hour after the lumbar medial branch block.

SECONDARY OUTCOMES:
Duration of low back pain | Baseline
  Participant self-reports the number of years they have experienced low back pain. The number of years for each participant will be reported.
PEG: A Three-Item Scale Assessing Pain Intensity and Interference | Baseline
  Assessment for self-reported average pain and pain interference within past 7 days. Responses range from 0 (no pain) to 10 (pain as bad as you can imagine). Total scores range from 0-30, and higher scores indicate more pain interference.
Baseline Back Pain Intensity | Baseline
  Assessment for determining how much a person hurts with a question ranked on a 11-point scale, from "0 = no pain" to "10 = worst imaginable pain." The minimum raw summed score is 0 and the maximum score is 10. Lower raw response scores suggest lower pain intensity and better outcomes.
PROMIS Pain Interference 4a | Baseline
  Assessment for self-reported consequences of pain with 4 questions ranked on a 5-point scale, from "not at all" to "very much". The minimum raw summed score is 4 and the maximum score is 20. Lower scores suggest better outcomes.
PROMIS Physical Function- 6b | Baseline
  Assessment for self-reported capability with 6 qualitatively scaled questions ranked on a 5-point scale, from "without any difficulty" to "unable to do" or "not at all" to "cannot do." The minimum raw summed score is 6 and the maximum score is 30.
PROMIS Sleep Disturbance 6a | Baseline
  Assessment for self-reported perceptions of sleep quality and sleep depth with 6 questions ranked on a 5-point scale. The minimum raw summed score is 6 and the maximum score is 30. Lower scores suggest better outcomes.
6-item Pain Catastrophizing Scale | Baseline
  Standardized survey score assessing pain perception before the study procedures begin. Rumination subscale score ranges from 0-16. Magnification subscale score ranges 0-12. Helplessness subscale score ranges from 0-24. Total score can be calculated by summing subscales. Total score ranges from 0-52, with higher scores indicating more pain catastrophizing.
Patient Health Questionnaire (PHQ-2) | Baseline
  The PHQ-2 inquires about the frequency of depressed mood and anhedonia over the past two weeks. The PHQ-2 includes the first two items of the PHQ-9. A PHQ-2 score ranges from 0-6. The authors identified a score of 3 as the optimal cutpoint when using the PHQ-2 to screen for depression.
  If the score is 3 or greater, major depressive disorder is likely.
PROMIS 4-item Depression | Baseline
  Assessment for self-reported negative mood and views of self with 4 questions ranked on a 5-point scale, from "never" to "always". The minimum raw summed score is 4 and the maximum score is 20. Lower t-scores suggest better outcomes.
PROMIS 4-item Anxiety | Baseline
  Assessment for self-reported fear, anxious misery, hyperarousal, and somatic symptoms with 4 questions ranked on a 5-point scale, from "never" to "always". The minimum raw summed score is 4 and the maximum score is 20. Lower scores suggest better outcomes.
Areas of Pain Body Map | Baseline
  The digital body figure contains 36 anterior regions and 38 posterior regions on which participants can mark areas in which they experience chronic pain. The number of pain areas each participant recorded will be reported, with a possibility of 74 total regions.
Treatment Expectancy | Baseline
  Assessment for the subject's expectations of treatment effec prior to lumbar medial branch block. Scores range from 0 (not at all) to 4 (very much), with total scores ranging from 0-24. Higher scores indicate higher expectations of the low back pain treatement.
Patient Global Impression of Change | Immediately after lumbar medial branch block
  The subject's impression of the impact of the lumbar medial branch block on their pain and function will be measured with a 7-item scale (1 = very much worse, 2 = much worse, 3 = minimally worse, 4 = no change, 5 = minimally improved, 6 = much improved, 7 = very much improved).
Situational pain catastrophizing scale (S-PCS) | Immediately after lumbar medial branch block
  Standardized survey score assessing pain perception immediately following the lumbar medial branch block. Scores range from 0-24, with higher scores representing more pain catastrophizing.
Pain intensity during QST | during this portion of the study visit (60 minutes)
  Changes in pain intensity during quantitative sensory tests measured on a 0-100 sliding scale (0 is no pain, 100 is the most intense pain imaginable)
Baseline back pain intensity | baseline
  Patients respond to the question "How would you rate your back pain on average?" from 0 (no pain) to 10 (worst imaginable pain) to see how intense their back pain is before the lumbar medial branch block.
Back pain intensity after lumbar medial branch block | Immediately after lumbar medial branch block and up to 16 hours after lumbar medial branch block
  Patients respond to the question "How would you rate your back pain right now?" from 0 (no pain) to 10 (worst imaginable pain) to see how intense their back pain is each hour after the lumbar medial branch block.

CONTACTS AND LOCATIONS:
Overall Officials: Benedict J Alter, MD, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC St. Margaret, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be available, including data dictionaries, after publication per journal and funding protocols. The statistical analysis plan and analytic code will also be available per the same protocols.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will become available after publication per journal and funding entity protocols.
Access Criteria: Data will be made available by reasonable request and/or per journal and funding entity protocols.